CLINICAL TRIAL: NCT02346630
Title: The Effect of Combining Robotic-Assisted Therapy With Levodopa/Carbidopa in Chronic Post-Stroke Upper-Limb Hemiparesis
Brief Title: Combining Robotic-Assisted Therapy and Pharmacotherapy in Post-Stroke Rehabilitation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We didn't receive the expected funding to support the study.
Sponsor: Ross D. Zafonte, MD (Other)
Responsible Party: Sponsor-Investigator, Ross D. Zafonte, MD, Principal Investigator, Spaulding Rehabilitation Hospital
Organization: Spaulding Rehabilitation Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-P-002440
Record Dates: First submitted 2014-12-16; First posted 2015-01-27 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Levodopa / Carbidopa + Armeo (Active Comparator): Levodopa / Carbidopa drug 100/25 mg once a day for 3 weeks. Armeo Robotic Assisted Intensive Upper Extremity Therapy every weekday for 3 weeks.
  Interventions: Drug: Levodopa / Carbidopa; Device: Armeo
- Placebo + Armeo (Placebo Comparator): Placebo capsules daily for 3 weeks. Armeo Robotic Assisted Intensive Upper Extremity Therapy every weekday for 3 weeks.
  Interventions: Drug: Placebo; Device: Armeo

INTERVENTIONS:
Drug: Placebo — Placebo capsules daily for 3 weeks.
  Other Names: Negative control
  Arms: Placebo + Armeo
Drug: Levodopa / Carbidopa — Levodopa / Carbidopa drug 100/25 mg once a day for 3 weeks.
  Other Names: Sinemet
  Arms: Levodopa / Carbidopa + Armeo
Device: Armeo — Armeo Robotic Assisted Intensive Upper Extremity Therapy every weekday for 3 weeks.

SUMMARY:
Stroke is the leading cause of acquired long-term disability in adults in developed countries. Despite aggressive rehabilitation, lasting upper extremity impairment remains in the majority of stroke survivors. It is hypothesized that enhancing neuroplasticity through the combination of drug therapy and physical therapy could enhance outcomes for stroke survivors. The combination of levodopa and intensive physical therapy shows promise in enhancing the functional motor recovery of stroke patients during the sub-acute and chronic period without reported significant side effects. Robotic-aided training is a promising tool that has the potential to deliver high-intensity, task-oriented, reproducible therapy that can decrease the burden on a therapist. Since the evidence behind dopaminergic potentiation of neuroplasticity and stroke recovery is promising, it is the investigators aim to combine dopaminergic drug therapy with highly intensive robotic-assisted therapy to provide superior upper extremity functional recovery over traditional stroke rehabilitation.

DETAILED DESCRIPTION:
Every year, approximately 795,000 people suffer a new or recurrent stroke in the United States, meaning that every 40 seconds someone has a stroke. In the United States, stroke is the third most frequent cause of death and the leading cause of lasting hemiparesis and adult disability. Since the prevalence of stroke increases with age, and since the world population is aging, the incidence of stroke is expected to rise in the coming years. This will become a significant societal burden since the care of stroke survivors is costly, to the individual and to society.

Post-stroke upper extremity (UE) impairment usually implies initial weakness, with subsequent diminished dexterity and limitation or incapacity for reaching, transport and grasping movements since the onset. Survivors may regain partial or, less often, complete muscle strength in the affected UE during the recovery process. However, a persistent degree of weakness and evolution to secondary complications as spasticity (characterized by increased flexor hypertonia), shoulder pain and contractures is frequent. These additional issues are associated with greater impairment, worse function and lower health-related quality of life. Treatment interventions for hemiparesis after stroke usually include stretching, strengthening of antagonist muscles, splinting, oral medications, and focal injections (phenol or botulinum toxin) and intrathecal baclofen. However, the amount, intensity and length of therapies still need further investigation. Despite adequate traditional treatment, a high number of patients are still permanently limited as a consequence of stroke. Based on motor learning theories, recent studies have demonstrated that intensive, repetitive, task-oriented therapies can help the paretic extremity "relearn" how to perform movements that were lost after brain damage.

ROBOTIC-ASSISTED UPPER-LIMB TRAINING WITH ARMEO®

Current evidence has shown that rehabilitation without specific training will not result in measurable outcomes. Factors such as intensity and specificity of motor training are important to achieve recovery of motor function, especially in the chronic phase of the stroke. There is robust evidence that highly-repetitive movement rehabilitation could improve motor and functional ability, based on its role in motor learning processes.Robotic devices have become a very important area of research because of their capacity to achieve high-intensity and specificity therapies.

In this proposed project, we plan to use the Armeo robotic system to deliver motor training therapy. The Armeo system is an adjustable arm orthosis that has received FDA 510k exemption. It passively counterbalances the weight of the arm, thereby reducing the effort required by the paretic arm to overcome gravity. The device is able to augment feedback through a virtual environment (i.e. computer games). The tasks presented in the virtual environment are designed to achieve functional movements, i.e. the subject has to perform tasks such as reaching for objects as part of the game. Gravity compensation, which can reduce the level of difficulty of performing an activity, facilitates active arm movement, especially when it involves training in grasping and reaching. By using the Armeo system, we hope to achieve repetitive training of reach, grasp, and release in an engaging environment that can be adapted to individual capabilities. We also expect to enable stroke survivors whose motor weakness may have excluded them from performing repetitive therapy tasks to participate in this study.

LEVODOPA Several agents have widely proved their influence on neuronal plasticity. Among these agents, pharmacological drugs increasing the availability of Central Nervous System (CNS) neurotransmitters (dopamine, norepinephrine, serotonin, acetylcholine and hista mine) have shown the ability to modulate excitability in cortical neurons and exert a subsequent facilitator effect in neuroplasticity. In this regard, several studies have been conducted in the past two decades investigating, among other agents, the effects of amphetamines, selective serotonin reuptake inhibitors, donepezil, psychostimulants as methylphenidate and dopaminergic agents. Levodopa (LD) is a desirable drug to evaluate because of its safe action profile. This oral medication is a precursor of dopamine (DA) that is actively transported across the blood-brain barrier and is converted to DA in the CNS and peripheral tissues. Approximately 95% of LD is converted to DA, stimulating dopaminergic neurotransmission, and the remaining 5% is converted to norepinephrine and affects adrenergic neurotransmission. DA plays a role in the formation of motor memories and thereby facilitates neuroplasticity, through the strengthening (long term potentiation, LTP) or weakening (long term depression, LTD) of the neuronal synapses, thereby generating neuroplasticity. DA has an inverted U-shape concentration curve effect to facilitate LTP. In previous studies doses of 100mg generated a facilitator effect, and 25 mg and 200 mg exerted an inhibitor effect on human cortex. This pharmacological agent has shown promising results in the treatment of stroke by enhancing functional motor recovery in the sub-acute and chronic period, in combination with intensive physical therapy, without reported significant side effects. In the acute and sub-acute phases, LD was demonstrated to improve functional motor skills that were maintained at three weeks follow up. LD also showed an additional benefit on the activities of daily living and in the severity of the stroke. In the chronic period, a single dose of LD combined with physical therapy for five weeks enhanced the formation of training-dependent elementary motor memory while improving UE dexterity.

COMBINING LEVODOPA/CARBIDOPA WITH THE ARMEO SYSTEM

It is our hypothesis that the intake of levodopa/carbidopa LD/CD in combination with intensive robotic-assisted therapy will provide better outcomes in functional recovery tests than the same training alone. We also hypothesize that these improvements could be correlated with changes in motor cortex excitability. Current strategies to improve motor recovery after stroke focus on neuroplasticity and neuromodulation. There is growing interest in the combination of therapies and strategies to enhance plasticity and thereby functional recovery through the rehabilitation process. It is frequently hypothesized that the combination of drug therapy and physical rehabilitation could provide better outcomes by enhancing neuroplasticity phenomenon

We propose a randomized, double-blind, placebo-controlled study of LD/CD in combination with repetitive upper-extremity functional task-oriented and robotic-aided training.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, community dwelling, age 18-85.
* First episode of stroke.
* Diagnosis of chronic ischemic stroke at least six months before study enrollment resulting in objective motor upper-extremity impairment as demonstrated during physical/neurological examination.
* Score of 15-55 out of 66 on the arm motor Fugl-Meyer scale.
* The ability to extend ≥ 10 degrees at metacarpophalangeal and interphalangeal joint of all digits.
* Signed written informed consent.

Exclusion Criteria:

* Intracranial hemorrhages.
* Pregnancy, planning to become pregnant or breast-feeding.
* History of seizures within the previous six months.
* Previous residual motor deficit in the affected side.
* Treatment with Botox injections in the affected arm in the previous 6 months.
* Cognitive impairment that may interfere with understanding instructions for motor tasks and assessment tools.
* Other major neurologic disorder (Parkinson's disease).
* Major depression defined by the Patient Health Questionnaire, other major psychiatric pathology, dementia, agitation (defined as a score of >21 on the Agitated Behavior Scale) or another uncooperative behavior.
* Inability to operate the Armeo system (which will be assessed during the calibration process). Subjects must have sufficient range of movement to enable calibration of the virtual workspace.
* Contraindications for Levodopa/ Carbidopa:

  * Hypersensitivity to levodopa, carbidopa or any component of the formulation.
  * Use of monoamine oxidase inhibitors (MAOIs) within prior 14 days. Treatment with tricyclic antidepressants, antipsychotics, sapropterin, selective serotonin reuptake inhibitors (SSRIs), pimozide, benzodiazepines, amantadine, methylphenidate, dopamine-agonists or neuroleptic drugs when inclusion or the month before.
  * Narrow-angle glaucoma.
  * Suspicious, undiagnosed skin lesions or a history of melanoma.
* Presence of metallic hardware in close contact to the discharging coil (cochlear implants, aneurism clips, brain implants, internal pulse generator, medication pumps).
* Contemporary participation in another interventional trial focused on the impaired arm recovery.
* Drug or alcohol abuse in the last 3 years.
* A terminal medical diagnosis with survival < 1 year.
* End-stage or uncompensated hepatic, cardiovascular, cerebrovascular, endocrine, renal, digestive, hematologic or pulmonary disease. Active ulcer disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Estimated); Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in Upper Extremity Score of the Fugl-Meyer Assessment (FM-UE) at 1 month | month 1
  FM-UE is an ordinal scale with scores ranging from 0 to 66 for upper-limb motor performance. It is composed of 33 items. FM-UE is a measure of upper-extremity motor impairment including coordination and speed.

SECONDARY OUTCOMES:
Computer Measures on the Armeo Robot | month 1
  Speed, movement accuracy and efficiency
Analysis of Muscle Activation Patterns During Upper Extremity Movements | month 1
  Electromyography Camera-based motion analysis
Transcranial Magnetic Stimulation Assessment (TMS) | month 1
  TMS is a non-invasive and non-painful method to evaluate changes in cortical brain excitability, which has been used in several studies in recent years to assess the response of pharmacological and non-pharmacological therapies in stroke survival patients.
Veteran's Rand 36 | month 1
  This is a generic health-related quality of life assessment comprised of 36 items.
Hand Dynamometry | month 1
  We will measure the grip strength of both hands using the Jamar® Hand Dynamometer. The time required is estimated to be less than 1 minute per hand.
Physical Examination | week 1
  Arm range of motion and muscle strength (Manual Muscle Testing).
Modified Ashworth Scale | month 1
  This scale represents a clinical measure of muscle spasticity.
Wolf Motor Function Test (WMFT) | month 1
  WMFT consists of 17 items that are UE motor tasks that can assess movement components required for daily tasks. Tasks are sequenced to progressively use more upper-extremity joints and include movements that range from simple patterns of motion to complex ones. Performance time, strength and quality of motor function are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Zafonte, DO, Principal Investigator — Harvard Medical School (HMS and HSDM); Paolo Bonato, PhD, Study Chair — Spaulding Rehabilitation Hospital; Duc A Tran, MD PhD, Study Director — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD